CLINICAL TRIAL: NCT03180879
Title: An Open Label, Randomised, Single Dose, Three-way Crossover Study to Compare the Bioavailability of 400 mg Ibuprofen From 2 x 200 mg Ibuprofen Acid Orodispersable Tablets, 2x 200 mg Ibuprofen Acid Tablets and 2 x 342 mg Ibuprofen Lysine Tablets in Fasted Healthy Volunteers
Brief Title: Ibuprofen Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RB7-UK-1604
Record Dates: First submitted 2017-05-17; First posted 2017-06-08 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1 (Experimental): Treatment Order: Test, Reference, Comparator
  Interventions: Drug: Test - RB ibuprofen acid orodispersible tablets; Drug: Reference - RB Nurofen ibuprofen acid tablets; Drug: Comparator - Dolormin ibuprofen lysine tablets
- 2 (Experimental): Treatment Order: Test, Comparator, Reference
  Interventions: Drug: Test - RB ibuprofen acid orodispersible tablets; Drug: Reference - RB Nurofen ibuprofen acid tablets; Drug: Comparator - Dolormin ibuprofen lysine tablets
- 3 (Experimental): Treatment Order: Reference, Test, Comparator
  Interventions: Drug: Test - RB ibuprofen acid orodispersible tablets; Drug: Reference - RB Nurofen ibuprofen acid tablets; Drug: Comparator - Dolormin ibuprofen lysine tablets
- 4 (Experimental): Treatment Order: Reference, Comparator, Test
  Interventions: Drug: Test - RB ibuprofen acid orodispersible tablets; Drug: Reference - RB Nurofen ibuprofen acid tablets; Drug: Comparator - Dolormin ibuprofen lysine tablets
- 5 (Experimental): Treatment Order: Comparator, Test, Reference
  Interventions: Drug: Test - RB ibuprofen acid orodispersible tablets; Drug: Reference - RB Nurofen ibuprofen acid tablets; Drug: Comparator - Dolormin ibuprofen lysine tablets
- 6 (Experimental): Treatment Order: Comparator, Reference, Test
  Interventions: Drug: Test - RB ibuprofen acid orodispersible tablets; Drug: Reference - RB Nurofen ibuprofen acid tablets; Drug: Comparator - Dolormin ibuprofen lysine tablets

INTERVENTIONS:
Drug: Test - RB ibuprofen acid orodispersible tablets — RB ibuprofen acid orodispersible tablets, 2 x 200 mg, single dose, oral.
Drug: Reference - RB Nurofen ibuprofen acid tablets — RB Nurofen ibuprofen acid tablets, 2 x 200 mg, single dose, oral.
Drug: Comparator - Dolormin ibuprofen lysine tablets — Dolormin ibuprofen lysine tablets 2 x 342 mg (each 342 mg tablet contains 200 mg ibuprofen), single dose, oral.

SUMMARY:
This project is the in-house development of a 200 mg ibuprofen acid orodispersable tablet (ODT; meltlet). It is designed to appeal to consumers who want a dosage form that may be taken without water and can be used 'on the go'. Vanquish has an improved organoleptic profile compared to the currently marketed meltet by the Sponsor. ODTs are also considered as a suitable dosage form for children who may be reluctant to swallow tablets. This product has the potential for application in both adults and children due to the convenience of the format and the ease of administration for both groups.

This will be the first pharmacokinetic (PK) assessment of the ibuprofen acid ODT formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who have given written informed consent.
2. Age: ≥ 18 years ≤ 50 years.
3. Body Mass Index (BMI) of ≥ 18.0 and ≤ 30 kg/m2.
4. Healthy as determined by past medical history, physical examination, vital signs, electrocardiogram (ECG), and laboratory tests at screening.
5. Female subject of child bearing potential with a negative pregnancy test at the screening visit and willing to use an effective method of contraception unless of non-childbearing potential or where abstaining from sexual intercourse in line with the preferred and usual lifestyle of the subject from first dose until 3 months after the final dose of study medication.
6. Female subject of non-child bearing potential with negative pregnancy test at the screening visit.
7. Male subject willing to use an effective method of contraception unless anatomically sterile or where abstaining from sexual intercourse in line with the preferred and usual lifestyle of the subject from first dose until 3 months after the final dose of study medication.

Exclusion Criteria:

1. Pregnant or lactating females.
2. A history and/or presence of significant disease of any body system, including significant psychiatric disorders, parasuicide.
3. Any condition that may currently interfere with the absorption, distribution, metabolism or excretion of drugs.
4. A history of allergy or intolerance related to treatment with ibuprofen, aspirin or other non-steriodal anti-inflammatory drugs (NSAIDs), or the excipients of the formulations
5. A history of or active peptic or duodenal ulcers or gastrointestinal bleed or upper gastro-intestinal bleed, or other significant gastro-intestinal disorders.
6. A history of frequent dyspepsia, e.g. heartburn or indigestion.
7. A history of significant and frequent migraine.
8. Current smokers or ex-smokers who have smoked or used nicotine replacement products during the 6 months prior to the first dose of study medication.
9. A history of substance abuse (including alcohol).
10. Consumption of foods or beverages containing caffeine (e.g. coffee, tea, cola and chocolate) above 300 mg caffeine per day, prior to 48 hours of each treatment period. (One cup of coffee equals approximately 50 mg caffeine).
11. Those with positive test for drugs of abuse and alcohol.
12. Ingestion of a prescribed drug at any time in the 14 days before the first dose of study medication (excluding hormonal contraceptives and hormone replacement therapy), or consumption of enzyme inhibitors or inducers 30 days prior to the first dose of study medication (such as barbiturates, carbamazepine, erythromycin, phenytoin, etc.).
13. Ingestion of an over-the-counter preparation within 7 days before the first dose of study medication, including herbal medications, vitamins, fish oil supplements, ibuprofen and other NSAIDs.
14. Those who have consumed grapefruit or grapefruit juice, pumelo or Seville oranges in the 7 days before the first dose of study medication.
15. Donation of blood > 400 mL e.g. to the blood transfusion service in the 12 weeks prior to the first dose of study medication.
16. Known human immune deficiency virus (HIV) positive status, or a positive viral serology test.
17. Topical use of ibuprofen within 7 days before the first dose of study medication.
18. Strenuous physical exercise from 48 hours prior to first dose of study medication.
19. Those previously randomised into this study.
20. Those who are an employee at the study site.
21. Those who are a partner or first degree relative of the Investigator.
22. Participation in a New Chemical Entity clinical study within the previous 3 months or a marketed drug clinical study within the 30 days before the first dose of study medication.
23. Those unable in the opinion of the Investigator to comply fully with the study requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
AUC0-t - the area under plasma concentration curve from administration to last quantifiable concentration at time t. | PK Analysis 0-12hrs
  The Test and Reference will be considered similar if for ibuprofen, for each corresponding PK parameter, the 90% confidence interval for the Test to Reference ratio (rounded to two decimal places) of LS geometric means is fully contained within the interval 80.00 to 125.00%:
Cmax - the maximum observed plasma concentration. | PK Analysis 0-12hrs
  The Test and Reference will be considered similar if for ibuprofen, for each corresponding PK parameter, the 90% confidence interval for the Test to Reference ratio (rounded to two decimal places) of LS geometric means is fully contained within the interval 80.00 to 125.00%:

SECONDARY OUTCOMES:
AUC0-t - the area under plasma concentration curve from administration to last quantifiable concentration at time t. | PK Analysis 0-12hrs
  The Test and Comparator will be considered similar if for ibuprofen, for each corresponding PK parameter, the 90% confidence interval for the Test to Comparator ratio (rounded to two decimal places) of LS geometric means is fully contained within the interval 80.00 to 125.00%:
Cmax - the maximum observed plasma concentration. | PK Analysis 0-12hrs
  The Test and Comparator will be considered similar if for ibuprofen, for each corresponding PK parameter, the 90% confidence interval for the Test to Comparator ratio (rounded to two decimal places) of LS geometric means is fully contained within the interval 80.00 to 125.00%:
Kel - Elimination rate constant | PK Analysis 0-12hrs
  Secondary endpoint for Test, Reference and Comparator products
AUC0-inf - Area under the plasma concentration-time curve from administration to infinity | PK Analysis 0-12hrs
  Secondary endpoint for Test, Reference and Comparator products
AUCR - Ratio AUC0-t/AUC0-inf | PK Analysis 0-12hrs
  Secondary endpoint for Test, Reference and Comparator products
Tmax - Time until Cmax is first achieved | PK Analysis 0-12hrs
  Secondary endpoint for Test, Reference and Comparator products
T1/2 - Plasma concentration (elimination) half-life | PK Analysis 0-12hrs
  Secondary endpoint for Test, Reference and Comparator products
Cn - The plasma concentration at each planned nominal time point. | PK Analysis 0-12hrs
  Secondary endpoint for Test, Reference and Comparator products

OTHER OUTCOMES:
Overall proportion of subjects with adverse events (AEs), i.e. the occurrence of one or more AEs per subject | Through study completion - Screening to study follow-up (approx 6 weeks)
Change from baseline in oral temperature. | Through study completion - Screening to study follow-up (approx 6 weeks)
  Measured in degrees Celcius
Change from baseline in resting heart rate. | Through study completion - Screening to study follow-up (approx 6 weeks)
  Measured in beats per minute
Change from baseline in resting blood pressure.. | Through study completion - Screening to study follow-up (approx 6 weeks)
  Measured in mmHg
Change from baseline in standard haematology testing. | Through study completion - Screening to study follow-up (approx 6 weeks)
Change from baseline in standard biochemistry testing. | Through study completion - Screening to study follow-up (approx 6 weeks)
Change from baseline in standard urinary testing. | Through study completion - Screening to study follow-up (approx 6 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Annelize Koch, MBBS, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research, Merthyr Tydfil, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sugar D, Francombe D, da Silva T, Hanid S, Hutchings S. Comparative Bioavailability Study of a New Orodispersible Formulation of Ibuprofen Versus Two Existing Oral Tablet Formulations in Healthy Male and Female Volunteers. Clin Ther. 2019 Aug;41(8):1486-1498. doi: 10.1016/j.clinthera.2019.04.040. Epub 2019 Jun 12. PMID 31202508